CLINICAL TRIAL: NCT06116058
Title: Integrated Neuromuscular Inhibition Technique Versus Instrument Assisted Soft Tissue Mobilization in Patients With Chronic Non Specific Low Back Pain
Brief Title: Integrated Neuromuscular Inhibition Versus Instrument Assisted Soft Tissue Mobilization in Chronic Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Salama Mansour Mousa, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004714
Record Dates: First submitted 2023-10-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Chronic Non Specific Low Back Pain
Keywords: chronic non specific low back pain; integrated nouromuscular inhibition technique; instrument assisted soft tissue mobilization technique
MeSH Terms: interventions — Methods; Exercise

STUDY DESIGN:
Intervention Model Description: 1. integrated neuromuscular inhibition technique and conventional physical therapy
  2. instrument assisted soft tissue mobilization technique and conventional physical therapy
  3. conventional physical therapy only
Who Masked: Participant, Outcomes Assessor
Masking Description: Double ( participant ,outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: integrated neuromuscular inhibition technique (Experimental): Group A: patient will receive integrated neuromuscular inhibition technique and conventional physical therapy program for 3 sessions /week over 4 weeks periods
  Interventions: Other: Experimental: Group A: integrated neuromuscular inhibition technique
- Group B :Instrument assissted soft tissue mobilization (Experimental): Group B : patient will receive Instrument assissted soft tissue mobilization technique and conventional physical therapy program for 3 sessions /week over 4 weeks periods
  Interventions: Other: Experimental: Group B :Instrument assissted soft tissue mobilization
- Group C:conventional physical therapy (Active Comparator): Group C: patient will receive conventional physical therapy only in the form of ( stretch for hamstring ,illiopoaps ,low back muscle and strenghtning for abdominal ,back muscles and side support exercise and quadriped exercise)
  Interventions: Other: control group C conventional physical therapy

INTERVENTIONS:
Other: Experimental: Group A: integrated neuromuscular inhibition technique — will receive integrated neuromuscular inhibition in addition to conventional treatment,INIT which included IC, SCS, and MET for the low back region for the quadratus lumborum( QL) and erector spinae (ES) muscles
  Other Names: technique
  Arms: Group A: integrated neuromuscular inhibition technique
Other: Experimental: Group B :Instrument assissted soft tissue mobilization — IASTM performed on lumbar posterior muscle erector spinae (iliocostalis, longissimus), and quadratus lumborum(QL) The IASTM treatment was applied for approximately 20-seconds in a direction parallel to the muscle fibers being treated with the instrument at a 45° angle. Followed immediately by treating the muscles in a direction perpendicular to the muscle fibers with the instrument at a 45° angle for an additional 20-seconds, resulting in a total treatment time of approximately 40 seconds.
  Other Names: instrument
  Arms: Group B :Instrument assissted soft tissue mobilization
Other: control group C conventional physical therapy — . The control group will applied general exercise. General exercise were applied with stretching exercises and stationary bicycling for 10-15 minutes14, 15) . Three sets of fifteen repetitions will performed, with rest times of 1 minute between sets during 4 weeks.
  Other Names: exercise
  Arms: Group C:conventional physical therapy

SUMMARY:
this study will be conducted to identify the difference between the effect of integrated neuromuscular inhibition technique and instrument assisted soft tissue mobilization on back pain, pain threshold, back rang of motion ,back proprioception and back disability in chronic non specific low back pain

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient's age ranged from 18 to 30 years.(Geogre et al, 2021) 2. Patients with low back pain for more than 3 months (pain felt between T12 and the gluteal fold).

  3. Patient with chronic low back pain 4. Normal body mass index from 18 -25kg/m2.

Exclusion Criteria:

* The subjects will be excluded if they have any of the followings:

  1. Lumbar discogenic lesions or any inflammatory arthritis, tumors, infection involving the lumbar spine.
  2. Patients with decreased range of motion secondary to congenital anomalies, muscular contracture, or bony block.
  3. Previous lumbar or hip surgery or trauma.
  4. Any hip structural abnormality such as malformations, impingements and degeneration.
  5. Patients With cognitive impairments that would limit their participation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
change in lumber proprioception | Evaluation will be performed priod to the first treatment session :as a baseline measure,and at least treatment session (after 4 weeks)as a post-treatment measure
  change in lumbar proprioception will be measured by dual inclinometer for 3 group pre-and post-treatment
chang in pain pressure threshold | Evaluation will be performed priod to the first treatment session :as a baseline measure,and at least treatment session (after 4 weeks)as a post-treatment measure
  change in lower back pain threshold will be measured by pressure algometer for 3 group pre-and post-treatment

SECONDARY OUTCOMES:
chang in lumbar rang of motion(ROM) | Evaluation will be performed priod to the first treatment session :as a baseline measure,and at least treatment session (after 4 weeks)as a post-treatment measure
  lumbar ROM will be measured by dual inclinometer pre-treatment and post treatment
functional disability oFlumbar spine | Evaluation will be performed priod to the first treatment session :as a baseline measure,and at least treatment session (after 4 weeks)as a post-treatment measure
  functional disability will be measured by The Arabic version of Oswestry Disability Index.(ODI)
pain level of lumbar spine | Evaluation will be performed priod to the first treatment session :as a baseline measure,and at least treatment session (after 4 weeks)as a post-treatment measure
  pain level will be measured by visual analoge scale(VAS)